CLINICAL TRIAL: NCT00039611
Title: Oxaliplatin (NSC 266046) in Combination With 5-Fluorouracil and Leucovorin (FOLFOX4) for Patients Who Have Not Received Prior Chemotherapy for Advanced Colorectal Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069434; CTEP-TRC-0201
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2002-07

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Clinical trial to study the effectiveness of combination chemotherapy in treating patients who have advanced colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Provide oxaliplatin in combination with fluorouracil and leucovorin calcium using the FOLFOX4 regimen for front-line treatment in patients with no prior chemotherapy for advanced colorectal cancer who are not eligible for entry into ongoing clinical trials of higher priority. (The regimen in this Treatment Referral Center protocol is one that was found to be superior in a recent national intergroup study.)
* Further determine the safety of this regimen in these patients.
* Further determine the anti-tumor activity of this regimen, defined as the rate of time-to-treatment failure, time to progression, and survival, in these patients.
* Capture data on subsequent salvage therapy administered to patients treated with this protocol.

OUTLINE: This is an open-label, multicenter study.

Patients receive oxaliplatin IV over 2 hours on day 1, leucovorin calcium IV over 2 hours on days 1 and 2, and fluorouracil IV over 22 hours on days 1 and 2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients with clinical evidence of benefit from this treatment, defined as stable disease, partial response, or complete response as well as no increase in size of any measurable or evaluable lesion and no new sites of disease, may be eligible for additional courses.

Patients are followed until death.

PROJECTED ACCRUAL: A maximum of 300 patients per month will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must not be eligible for Inter-group, Cooperative Group, or local clinical trials of higher priority
* Histologically or cytologically confirmed colorectal adenocarcinoma

  * Locally advanced or metastatic
  * Not curable by surgery or amenable to radiation therapy with curative intent
* Site of primary lesion must be or have been in the large bowel, as confirmed endoscopically, radiologically, or surgically
* No separate histological or cytological confirmation of metastatic disease is required for patients with a history of colorectal cancer treated by surgical resection who develop radiological or clinical evidence of metastatic cancer unless:

  * More than 5 years has elapsed since prior primary surgery and the development of metastatic disease OR
  * Primary cancer was a Duke's A or B1 lesion
* Measurable or evaluable disease
* No prior chemotherapy for advanced colorectal cancer

  * Prior adjuvant therapy allowed for resected stage II, III, or IV disease with any regimen containing fluorouracil with or without irinotecan or with immunotherapy, provided recurrent disease has been documented

PATIENT CHARACTERISTICS:

Age:

* 15 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL (transfusion allowed)

Hepatic:

* Bilirubin no greater than 1.5 mg/dL (regardless of liver involvement secondary to tumor)
* AST less than 5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No uncontrolled high blood pressure
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No myocardial infarction within the past 6 months
* No New York Heart Association class III-IV cardiac disease

Pulmonary:

* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* No pleural effusion or ascites that causes respiratory compromise (i.e., dyspnea grade 2 or greater)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions to compounds of similar chemical or biologic composition to platinum agents or oxaliplatin as well as other study agents
* No neuropathy grade 2 or greater, regardless of causality
* No HIV-positive patients receiving combination anti-retroviral therapy
* No ongoing or active infection
* No uncontrolled concurrent illness
* No psychiatric or social situations that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No concurrent sargramostim

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior major radiotherapy (e.g., chest or bone palliative radiotherapy)

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior major surgery (e.g., laparotomy)
* At least 2 weeks since prior minor surgery
* Insertion of a vascular access device is not considered major or minor surgery

Other:

* Recovered from effects of prior treatment
* No other concurrent investigational agents
* No oral cryotherapy on day 1 of each course

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-05; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Percy Ivy, MD, Study Chair — NCI - Investigational Drug Branch
Locations (19):
- United States (19):
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of California San Diego Cancer Center, La Jolla, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - Atlanta Cancer Care, Atlanta, Georgia
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - Cancer Therapy Evaluation Program, Bethesda, Maryland
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - St. Vincent Hospital and Health Center, Billings, Montana
  - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Ireland Cancer Center, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington